CLINICAL TRIAL: NCT02644057
Title: Comparison of Dobutamine Versus Milrinone for Renal Recovery in Patients With Cardiorenal Syndrome-A Prospective Cohort Study in Patients With Acute Decompensated Heart Failure
Brief Title: Dobutamaine Versus Milrinone in Cardiorenal Syndrome
Acronym: DOMICAS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not enroll patients
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Norbert Moskovits, Departmental head , Division of Heart Failure, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-05-11-MMC
Record Dates: First submitted 2015-10-29; First posted 2015-12-31 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-03

CONDITIONS: Cardiorenal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — Milrinone; Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- M-group (Active Comparator): Will be given milrinone as an intravenous infusion at 0.2-0.6 mcg/kg/min for a maximum period of 72 hours and adjusted based on creatinine clearance measured by cockcroft-gault equation. It would be titrated based on hemodynamic response , urine output and at the discretion of the treating physician
  Interventions: Drug: Milrinone
- D-group (Active Comparator): Will be given dobutamine as an intravenous infusion at a maximum rate of 20 mcg/kg/min depending on patient tolerance and would adjusted based on hemodynamic response, urine output and at the discretion of treating physician
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Milrinone — Patients who meet the inclusion criteria for the study will receive milrinone and patients will be monitored for improvement of the renal function objectively with measures such as Blood urea nitrogen, creatinine , daily urine output and changes in weight
  Arms: M-group
Drug: Dobutamine — Patients who meet the inclusion criteria for the study will receive dobutamine and patients will be monitored for improvement of the renal function objectively with measures such as Blood urea nitrogen, creatinine , daily urine output and changes in weight
  Arms: D-group

SUMMARY:
Heart failure is recognized as one of the most common indications for hospitalization amongst adults aged >65 years in United States with estimated Medicare cost to be 17 billion or more. Chronic heart failure is one of the most life threatening cardiovascular disorder thought to affect nearly six million US population with 600,000 new cases every year. The heart is responsible for perfusion to all vital organs including kidneys and dysfunction in either affects both the vital organs. When dysfunction of heart leads to dysfunction of kidneys or vice versa it is referred to as cardio renal syndrome (CRS). The underlying pathophysiology for CRS has been poorly understood and considered multifactorial. Worsening renal function defined as increase in serum creatinine of >0.3mg/dl from baseline occurs in 20-30% of patients with ADHF and is associated with greater length of hospital stay, hospital readmission and death. A number of interventions have been used including giving diuretics which helps in decongestion and helps the heart pump blood more effectively. Sometimes these therapies are not effective and may even lead to worsening of renal function. In such cases , inotrope agents which increase the contractility of the heart have been used to help pump more blood to vital organs. There have been very few trials assessing the efficacy of these agents for improving kidney function .The investigators aim to assess the renal recovery with two such agents - dobutamine and milrinone in patients with cardiorenal syndrome who are coming with acute decompensated heart failure

DETAILED DESCRIPTION:
Heart failure is recognized as one of the most common indications for hospitalization amongst adults aged >65 years in United States with estimated Medicare cost to be 17billion or more. Chronic heart failure is one of the most life threatening cardiovascular disorder thought to affect nearly six million US population with annual death rate being 600,000. Cardiorenal syndrome although not completely understood in its full context - is a term coined for disorder of the heart and kidneys whereby acute or chronic dysfunction of one precipitates acute or chronic dysfunction of the other. Concomitant kidney failure amongst patients with acute decompensated heart failure is commonly observed . Direct and indirect effects of heart failure other than hemodynamic insult have been identified as primers for acute kidney injury and dysfunction. Patients with preexisting underlying renal disease are more likely to develop worsening renal failure in the setting of ADHF with venous congestion being the most important hemodynamic factor driving it. Worsening renal function defined as increase in serum creatinine of >0.3mg/dl from baseline occurs in 20-30% of patients with ADHF and is associated with greater length of hospital stay, hospital readmission and death. The treatment of ADHF which includes the step up intravenous diuretic therapy in addition to optimizing baseline medicines is limited frequently by diuretic resistance and worsening creatinine level precluding use of Angiotensin converting enzyme inhibitors (ACEi), Angiotensin Receptor Blocking Agents (ARBs), and Spironolactone. Ultrafiltration/Aquapheresis still remains an option for treating non-responders to medical therapy. Inotropes have been known to produce a beneficial hemodynamic effect on heart and lead to better titration to oral regimen. Short term continous intravenous infusion of inotropic agents in patients with documented severe systolic dysfunction who present with significantly depressed cardiac output to maintain end organ perfusion has been shown to be beneficial as per the ACC/AHA guidelines 2013 for management of heart failure. The use of intravenous inotropes remains still a controversial topic in terms of its short lived and long term efficacy on renal recovery in acute decompensated heart failure. In view of the large proportion of patients admitted with acute decompensated heart failure and no real world studies comparing different inotropes to improve kidney function, the investigators aim to compare the efficacy of dobutamine and milrinone in improving kidney function and also their effect on length of stay, symptomatic improvement and medication optimisation

1. The primary objective of the study is to objectively measure the response of dobutamine vs milrinone for renal recovery in patients with cardiorenal syndrome (>0.3mg/dl increase in creatinine from baseline) admitted for acute decompensated heart failure. These objective measures include change in serum creatinine, change in weight.
2. The secondary objectives are to measure the length of hospitalization, readmission rates and unscheduled visits to the clinic or ER during 60 day follow up period. The investigators will also measure changes in symptoms which will be assessed using global and dyspnea visual analog scale every 24 hours until the patient is discharged .
3. The secondary objectives also include to measure diuretic dose, medicine optimization including initiation of beta blocker / ace inhibitors before discharge, at 30 days and 60 days interval
4. The investigators will subdivide the patients into ischemic versus non ischemic at the end of trial to see the response in both these categories of patients

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Admitted to the hospital with a primary diagnosis of Decompensated Heart Failure
3. Onset of cardio-renal syndrome (increasing creatinine>0.3mg/dl) after or before hospitalization. After hospitalization within 7 days of from the time of admission after receiving intravenous diuretics and heart failure medication optimization. Before hospitalization in the setting of escalating doses of outpatient loop diuretics and heart failure medication optimization
4. Persistent volume overload- For patients with a pulmonary artery catheter, peristent volume overload will include :

   Pulmonary capillary wedge pressure >22mm Hg and one of the following clinical signs :2+ peripheral edema and/or pulmonary edema or pleural effusion on chest Xray. For patients without a pulmonary artery catheter- persistent volume overload will include atleast 2 of the following: 2+ peripheral edema , jugular venous pressure >10 mm Hg and pulmonary edema or pleural effusion on chest Xray
5. BNP>400
6. Cr-1.2-3.0

Exclusion Criteria:

1. Intravascular volume depletion
2. Acute coronary syndrome within 4 weeks
3. Indication for hemodialysis
4. Systolic Blood pressure <90mm Hg or MAP<60mm Hg at the time of enrollment
5. Alternate explanation for worsening renal function , such as obstructive nephropathy , contrast induced nephropathy , ATN
6. Clinical instability likely to require the addition of intravenous vasoactive drugs including vasodilators and/or inotropic drugs
7. The use of iodinated radio-contrast material in the past 72 hours or anticipated use of intravenous contrast during the current hospitalization
8. Underlying rhythm disorder

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Estimated); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Serum creatinine measured in mg/dl(milligram/decilitre) | Serum Creatinine would be measured every 24 hours in mg/dl from the time of enrollment in the study and will be measured every 24 hours up to a maximum period of 14 days

SECONDARY OUTCOMES:
Length of hospitalisation | Length of stay measured in days up to a maximum of 30 days
  Length of stay will start from the day patient is admitted up to a maximum of 30 days
Readmission rate | Readmissions would be assessed for a period of 90 days
Global visual analog score | Every 24 hours from the day of enrollment in the study up to a maximum period of 14 days
Dyspnea visual analog score | Every 24 hours starting from the day of enrollment in the study up to a maximum period of 14 days
Urine output measured in milliliters in a 24 hour period | Every 24 hours from the day of enrollment in the study up to a maximum period of 14 days
  Urine output would be strictly monitored in millilitres /24 hours starting from the day of enrollment in the study till the patient is discharged from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Moskovits, MD, Principal Investigator — Maimonides Medical Center; Karan Wats, MBBS, Principal Investigator — Maimonides Medical Center; Syeda A Batul, MBBS, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Ronco C, Haapio M, House AA, Anavekar N, Bellomo R. Cardiorenal syndrome. J Am Coll Cardiol. 2008 Nov 4;52(19):1527-39. doi: 10.1016/j.jacc.2008.07.051. PMID 19007588
- [Background] Abraham WT, Adams KF, Fonarow GC, Costanzo MR, Berkowitz RL, LeJemtel TH, Cheng ML, Wynne J; ADHERE Scientific Advisory Committee and Investigators; ADHERE Study Group. In-hospital mortality in patients with acute decompensated heart failure requiring intravenous vasoactive medications: an analysis from the Acute Decompensated Heart Failure National Registry (ADHERE). J Am Coll Cardiol. 2005 Jul 5;46(1):57-64. doi: 10.1016/j.jacc.2005.03.051. PMID 15992636
- [Background] Cuffe MS, Califf RM, Adams KF Jr, Benza R, Bourge R, Colucci WS, Massie BM, O'Connor CM, Pina I, Quigg R, Silver MA, Gheorghiade M; Outcomes of a Prospective Trial of Intravenous Milrinone for Exacerbations of Chronic Heart Failure (OPTIME-CHF) Investigators. Short-term intravenous milrinone for acute exacerbation of chronic heart failure: a randomized controlled trial. JAMA. 2002 Mar 27;287(12):1541-7. doi: 10.1001/jama.287.12.1541. PMID 11911756
- [Background] Elkayam U, Tasissa G, Binanay C, Stevenson LW, Gheorghiade M, Warnica JW, Young JB, Rayburn BK, Rogers JG, DeMarco T, Leier CV. Use and impact of inotropes and vasodilator therapy in hospitalized patients with severe heart failure. Am Heart J. 2007 Jan;153(1):98-104. doi: 10.1016/j.ahj.2006.09.005. PMID 17174645